CLINICAL TRIAL: NCT05564780
Title: Study of Early Pharmaceutical Intervention for Cardiovascular Disease Prevention in Stage 1 Hypertension
Acronym: STEP-Pre
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Jun Cai, MD, PhD, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-GSP-GG-5
Record Dates: First submitted 2022-09-29; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Cardiovascular Diseases
Keywords: Stage 1 Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Antihypertensive drugs will be provided to the participants in the arm, including RASI and/or a single pill combination based on RASI.
  If the blood pressure of a participant elevates to above 140/90 mmHg, antihypertensive therapy will be provided.
  Interventions: Drug: RASI and/or a single pill combination based RASI
- Control (No Intervention): If the blood pressure of a participant elevates to above 140/90 mmHg, antihypertensive therapy will be provided.

INTERVENTIONS:
Drug: RASI and/or a single pill combination based RASI — The participants in the Treatment group will begin with a single category antihypertensive drug to control their blood pressure, for example, perindopril. If the blood pressure cannot be controlled under 130/80 mmHg, another type of antihypertensive drug will be added.
  Arms: Treatment

SUMMARY:
STEP-Pre is to investigate the benefits of using anti-hypertensive drugs in the population with a blood pressure of 130-139/80-89 mmHg and evaluate the health economics.

STEP-Pre is a multi-center randomized clinical trial. The cohort will be randomized into the treatment group or control group with a 1:1 ratio. The treatment group will take anti-hypertensive medicine to control blood pressure under 130/80 mmHg. Both groups will take health care education.

STEP-Pre will last 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Stage 1 hypertension (blood pressure is in 130-139/80-89 mmHg);
* 35 - 64 years old
* Without taking antihypertensive medicine during screening
* Signed the written informed consent

Exclusion Criteria:

* took antihypertensive medicine within the last 1 month;
* History of large atherosclerotic cerebral infarction or hemorrhagic stroke (not lacunar infarction and transient ischemic attack [TIA]);
* History of myocardial infarction or unstable angina or history of coronary revascularization (PCI or CABG);
* Lab tests indicating abnormal liver or kidney function (ALT ≥ 3 times the upper limit of normal value, or estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m2);
* History of sustained atrial fibrillation or Ventricular arrhythmias at entry influencing the measurement of electronic blood pressure；
* Severe valvular disease or valvular disease likely to require surgery or percutaneous valve replacement during the trial;
* Dilated or hypertrophic cardiomyopathy, rheumatic heart disease, or congenital heart disease;
* Severe somatic disease such as cancer;
* Severe cognitive impairment or mental disorders;
* pregnant or breastfeeding, or planning to be pregnant;
* having organ transplantation;
* Participating in other clinical trials.

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20000 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular Disease | 4 years
  A composite end-point comprised of acute coronary syndrome (myocardial infarction and hospitalization for unstable angina), first occurrence of symptomatic stroke ( ischemic or hemorrhagic stroke), and death from cardiovascular causes.

SECONDARY OUTCOMES:
Stroke ( ischemic or hemorrhagic) | 4 years
  Stroke is defined as a rapid onset of focal (or global) disturbance of cerebral function lasting more than 24 hours (except interrupted by surgery or death) without resolution of symptoms according to the World Health Organization. The diagnosis of stroke is confirmed by strict neurological examination, computed tomography (CT), or magnetic resonance imaging (MRI), and stroke subtypes are classified including ischemic or hemorrhagic, fatal or not fatal.
Acute coronary syndrome | 4 Years
  Acute coronary syndrome includes myocardial infarction and hospitalization for unstable angina. The diagnosis of MI is based on the following criteria: (1) Patient has cardiac signs and symptoms, such as retrosternal pain last for at least 30 minutes, and not relieve to nitroglycerine during the attack; (2) Electrocardiographic abnormal findings of MI are observed; (3) Biochemical markers of cardiac damage are present.
  The diagnosis of unstable angina requires hospitalization for evaluation. The clinical presentation of unstable angina includes: (1) prolonged (>20 min) angina pain at rest; (2) new onset angina; (3) post-MI angina; (4) recent destabilization of previously stable angina with at least Canadian Cardiovascular Society Class III angina characteristics.
CVD Death | 4 Years
  Cardiovascular death includes fatal coronary heart disease, fatal stroke, death from heart failure, and sudden cardiac death.
Advanced to Stage 2 Hypertension | 4 Years
  the proportion of participants with blood pressure increasing to above 140/90 mmHg.

IPD SHARING:
Plan to Share IPD: Yes
The collected data, study protocol, and SAP are planned to be shared after the study ends 5 years later.
Supporting Information: Study Protocol, SAP